CLINICAL TRIAL: NCT02325180
Title: Clinical Efficacy of Artemisinin-based Combination Therapy for Treatment of Uncomplicated Plasmodium Falciparum Malaria in North Sumatera, Indonesia and the Association of Molecular Markers With Treatment Outcomes
Brief Title: Artemisinin-based Combination Therapy for Treatment of Plasmodium Falciparum Malaria in North Sumatera, Indonesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Universitas Sumatera Utara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QA620
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Malaria, Falciparum
Keywords: ACT; Plasmodium falciparum; malaria; efficacy; Indonesia
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA-PQ (Experimental): One tablet of dihydroartemisinin-piperaquine consists of 40 mg of dihydroartemisinin and 320 mg of piperaquine. DHA-PQ is administered once daily for 3 days (at enrolment, hour 24 and you 48). Dosing should be given based on body weight. Daily dose for dihydroartemisinin is 2.25 mg/kg (total 6.75 mg/kg) and for piperaquine is 18 mg/kg (total 54 mg/kg).
  Interventions: Drug: Dihydroartemisinin-Piperaquine
- AL (Active Comparator): Half a tablet of artemether-lumefantrine consists of 20 mg of artemether and 120 mg of lumefantrine is given per 5 kg body weight. AL is administered as 6-dose regimens given twice daily for 3 days (at enrolment, hour 8, hour 24, hour 36, hour 48 and hour 60).
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine
  Other Names: Duo-Cotecxin; Artekin
  Arms: DHA-PQ
Drug: Artemether-lumefantrine
  Other Names: Coartem
  Arms: AL

SUMMARY:
This is a prospective, open label, randomised controlled trial to assess the safety and efficacy of dihydroartemisinin-piperaquine and artemether-lumefantrine in children and adults with uncomplicated Plasmodium falciparum malaria infection. Molecular markers for antimalarial resistance will also be assessed and the presence of molecular markers in the parasites will be associated with treatment outcomes.

DETAILED DESCRIPTION:
Artemisinin-based combination therapy (ACT) is the current recommended treatment by WHO for uncomplicated falciparum malaria. It is highly effective with few adverse effects. The artemisinin component is combined with a partner drug with a longer half-life to ensure the clearance of the remaining parasites after rapid reduction by artemisinin.

ACT is used as first-line treatment for uncomplicated P. falciparum infection in Indonesia since 2004. There are 3 combinations available in the country including artesunate-amodiaquine (AS-AQ), dihydroartemisinin-piperaquine (DHA-PQ) and artemether-lumefantrine (AL). Studies at different sites across Indonesia have shown various efficacy. Yet, there is an increased concern of reduced susceptibility of P. falciparum to artemisinin in neighbouring countries. Therefore, there is a need to evaluate and monitor the efficacies of these combinations in Indonesia.

Molecular markers are an important tool for detecting and monitoring the presence of antimalarial resistance. Their significant implication is to geographically map the extent of resistant-parasites, thus enabling strategies for their control and elimination to be applied before the inevitably increase in the disease burden occurs. Different markers have been used to identify antimalarial resistance and recently a molecular marker for artemisinin susceptibility in P. falciparum has also been proposed. The presence of these markers in parasites from our study will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* All patients per 6 months of age
* Fever as defined by axillary temperature > 37.5 C or history of fever during the 48 hours before recruitment
* Infection with P. falciparum detected by microscopy
* Parasitaemia > 250 /uL blood
* Ability to swallow oral medication
* Ability and willingness to comply with the protocol for the duration of the study and to comply with the study visit schedule
* Informed consent from the patient or from a parent or guardian in the case of children
* Absence of history to hypersensitive reactions or contraindication to antimalarial drugs
* Not currently consuming antibiotic with antimalarial activity (such as cotrimoxazole, macrolides, tetracycline or doxycycline)

Exclusion Criteria:

* Presence of general danger signs in children under 5 years or signs of severe falciparum malaria according to the definitions of WHO (2000)
* Presence of severe malnutrition according to WHO child growth standards
* Presence of febrile conditions caused by diseases other than malaria
* Presence of severe anemia (Hemoglobin < 7 gr/dL)
* Received any of the study drugs within the past 4 weeks
* Received any antimalarial within the last 2 weeks
* Recurrent vomiting )necessitating more than a single repeat dose)
* Pregnant (demonstrated by positive result of b-HCG in women of childbearing age
* Lactating mother

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of dihydroartemisinin-piperaquine and artemether-lumefantrine | 42 days
  Early treatment failure, late treatment failure, adequate clinical and parasitological response Proportion of participants with Adequate Clinical and Parasitological Response

SECONDARY OUTCOMES:
Parasite clearance times | 3 days
  Parasite reduction ratio, parasite clearance half-life
Fever clearance times | 3 days
Prevalence of molecular markers and the impact on treatment outcomes | 42 days
  Pfcrt, Pfmdr1, Pfk13 and any other important molecular markers
Prevalence of gametocyte | 42 days
  Proportion of patients with gametocyte
Presence of other Plasmodium species | 42 days
  Plasmodium vivax, Plasmodium malariae, Plasmodium ovale spp, Plasmodium knowlesi
Haematological recovery | 28 days
  Haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Colin J Sutherland, BSc PhD MPH, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (3):
- Indonesia (3):
  - Primary health centres, Kuala Langkat, North Sumatera
  - Primary health centres, Tanjung Tiram, North Sumatera
  - Pulau-pulau Batu health centres, Tello Island, North Sumatera

REFERENCES:
- [Background] Guidelines for the Treatment of Malaria. 2nd edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK254223/ PMID 25473692
- [Background] White NJ, Pukrittayakamee S, Hien TT, Faiz MA, Mokuolu OA, Dondorp AM. Malaria. Lancet. 2014 Feb 22;383(9918):723-35. doi: 10.1016/S0140-6736(13)60024-0. Epub 2013 Aug 15. PMID 23953767
- [Background] Fairhurst RM, Nayyar GML, Breman JG, Hallett R, Vennerstrom JL, Duong S, Ringwald P, Wellems TE, Plowe CV, Dondorp AM. Artemisinin-resistant malaria: research challenges, opportunities, and public health implications. Am J Trop Med Hyg. 2012 Aug;87(2):231-241. doi: 10.4269/ajtmh.2012.12-0025. PMID 22855752
- [Background] Noedl H, Se Y, Schaecher K, Smith BL, Socheat D, Fukuda MM; Artemisinin Resistance in Cambodia 1 (ARC1) Study Consortium. Evidence of artemisinin-resistant malaria in western Cambodia. N Engl J Med. 2008 Dec 11;359(24):2619-20. doi: 10.1056/NEJMc0805011. Epub 2008 Dec 8. No abstract available. PMID 19064625
- [Background] Dondorp AM, Nosten F, Yi P, Das D, Phyo AP, Tarning J, Lwin KM, Ariey F, Hanpithakpong W, Lee SJ, Ringwald P, Silamut K, Imwong M, Chotivanich K, Lim P, Herdman T, An SS, Yeung S, Singhasivanon P, Day NP, Lindegardh N, Socheat D, White NJ. Artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2009 Jul 30;361(5):455-67. doi: 10.1056/NEJMoa0808859. PMID 19641202
- [Background] White NJ. Malaria: a molecular marker of artemisinin resistance. Lancet. 2014 Apr 26;383(9927):1439-1440. doi: 10.1016/S0140-6736(14)60656-5. No abstract available. PMID 24766952
- [Background] Ariey F, Witkowski B, Amaratunga C, Beghain J, Langlois AC, Khim N, Kim S, Duru V, Bouchier C, Ma L, Lim P, Leang R, Duong S, Sreng S, Suon S, Chuor CM, Bout DM, Menard S, Rogers WO, Genton B, Fandeur T, Miotto O, Ringwald P, Le Bras J, Berry A, Barale JC, Fairhurst RM, Benoit-Vical F, Mercereau-Puijalon O, Menard D. A molecular marker of artemisinin-resistant Plasmodium falciparum malaria. Nature. 2014 Jan 2;505(7481):50-5. doi: 10.1038/nature12876. Epub 2013 Dec 18. PMID 24352242
- [Derived] Lubis IND, Wijaya H, Lubis M, Lubis CP, Beshir KB, Staedke SG, Sutherland CJ. Recurrence of Plasmodium malariae and P. falciparum Following Treatment of Uncomplicated Malaria in North Sumatera With Dihydroartemisinin-Piperaquine or Artemether-Lumefantrine. Open Forum Infect Dis. 2020 Apr 2;7(5):ofaa116. doi: 10.1093/ofid/ofaa116. eCollection 2020 May. PMID 32420402